CLINICAL TRIAL: NCT07089433
Title: Morbidity Following Free Gingival Graft Harvesting With or Without the Use of the Palatal Shield Technique as a Wound Dressing: A Randomized Trial
Brief Title: Palatal Shield Technique for Graft Donor Site Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Palatal Shield
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Palatal Wound
Keywords: Free gingival graft; Wound healing; palatal stent
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): The palatal wound will be protected with composite resin
  Interventions: Procedure: Palatal stent as wound dressing
- Control (Active Comparator): The palatal wound will be covered with collagen sponge
  Interventions: Procedure: Conventional suturing

INTERVENTIONS:
Procedure: Palatal stent as wound dressing — The palatal wound after graft harvesting will be protected with a flowable composite resin adhesively secured to adjacent teeth
  Arms: Test
Procedure: Conventional suturing — The wound will be covered with a collagen sponge that will be hold in place with sutures
  Arms: Control

SUMMARY:
This randomized clinical trial aims to compare two techniques for managing the palatal donor site following gingival graft harvesting: a palatal stent made of flowable composite resin versus conventional suturing. The primary goal is to identify which method provides superior patient-reported outcomes (PROMs), thus optimizing postoperative comfort and overall patient well-being.

Systemically healthy patients, free of active periodontitis, requiring a palatal graft as part of periodontal or peri-implant mucogingival surgeries will be recruited and randomized into two groups. The experimental group will receive a palatal shield made of flowable composite resin adhesively secured to adjacent teeth, whereas the control group will undergo conventional suturing. In both groups, a collagen hemostatic sponge will be placed to aid hemostasis.

Primary endpoints include postoperative pain measured daily via Visual Analog Scale (VAS), general patient comfort during daily activities such as eating and oral hygiene, and overall patient satisfaction assessed using Likert scales or validated questionnaires.

Secondary endpoints involve clinical healing evaluated clinically and photographically at 7 and 14 days postoperatively, incidence of postoperative complications (e.g., prolonged bleeding, infections), analgesic consumption, functional recovery time, and oral health-related quality of life measured by the OHIP-14 questionnaire.

Statistical analysis will compare groups using appropriate parametric or non-parametric tests for continuous variables (pain scores, recovery time) and Chi-square or Fisher's exact tests for categorical variables. Pain progression over time will be assessed using repeated-measures ANOVA or an equivalent non-parametric test.

This study will help determine whether the palatal stent represents a superior alternative to conventional techniques in improving patient comfort, healing, and postoperative oral health-related quality of life in mucogingival surgical procedures.

DETAILED DESCRIPTION:
Objective This study aims to compare the effectiveness of palatal stent management versus conventional suturing on patient-reported outcome measures (PROMs), to identify the optimal strategy for managing palatal donor sites and improving postoperative patient well-being.

Primary Endpoints

* Postoperative Pain: Measured daily using a Visual Analog Scale (VAS) during the first postoperative week.
* General Patient Comfort: Evaluated using standardized questionnaires assessing discomfort during daily activities such as eating and oral hygiene.
* Patient Satisfaction: Assessed using Likert scales or validated questionnaires.

Secondary Endpoints

* Clinical Healing of Donor Site: Evaluated clinically (e.g., redness, swelling, infection signs) and photographically at 7 and 14 days postoperatively.
* Postoperative Complications: Frequency of events including prolonged bleeding, infection, or need for additional intervention.
* Analgesic Use: Number and duration of analgesic doses prescribed or voluntarily taken by patients.
* Functional Recovery Time: Days required for patients to resume normal activities (e.g., eating without difficulty, returning to work).
* Oral Health-Related Quality of Life: Evaluated using standardized questionnaires such as OHIP-14.

Study Design

Eligible patients will be recruited and randomized into two groups:

* Experimental Group: Palatal shield management using flowable composite resin secured by adhesion to the palatal surfaces of adjacent teeth.
* Control Group: Conventional suturing management.

Prior to the procedure, baseline clinical information including plaque index and bleeding index will be collected, and informed consent will be obtained from each patient.

Surgical Procedure Free gingival graft harvesting will be performed from the palate according to standard surgical techniques. The recipient surgical procedure is not within the scope of this study and will not influence the outcomes. In both groups, collagen sponge hemostatic dressing will be secured on the donor site using either resin or sutures.

Postoperative Care All patients will receive standardized postoperative instructions, including oral hygiene and pain management guidelines, along with analgesic prescriptions as needed. Follow-up evaluations will be conducted at 1 and 2 weeks postoperatively to assess pain (VAS), complications, and healing status. Patients will complete standardized questionnaires measuring comfort, satisfaction, and oral health-related quality of life.

Inclusion Criteria Systemically healthy patients without active periodontitis requiring periodontal or peri-implant mucogingival surgery involving palatal graft harvesting.

Independent Variables

* Donor Site Management Technique:
* Palatal stent (Experimental group)
* Conventional suture (Control group)

Dependent Variables

* Postoperative pain (VAS)
* Perceived comfort (standardized questionnaires)
* Clinical healing (clinical observations)
* Postoperative complications
* Analgesic consumption
* Functional recovery time
* Patient satisfaction
* Oral health-related quality of life (OHIP-14)

Confounding Variables

* Patient age
* Gender
* Smoking status
* Graft dimensions (width and depth)

Statistical Analysis Data will be analyzed using appropriate statistical methods to compare both groups. Continuous variables, such as pain scores and recovery time, will be analyzed using independent samples t-test or Mann-Whitney U test based on data distribution. Categorical variables, such as complications and analgesic use, will be evaluated using Chi-square or Fisher's exact test. Pain evolution over time will be assessed using repeated-measures ANOVA or non-parametric equivalents. Quality of life questionnaires (OHIP-14) and patient satisfaction scores will be analyzed using descriptive statistics and between-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) requiring periodontal or peri-implant mucogingival surgery involving palatal graft harvesting.
* Systemically healthy patients without medical conditions affecting wound healing.
* Patients free of active periodontal disease at the time of surgery.
* Patients able and willing to comply with postoperative instructions, complete questionnaires, and attend follow-up appointments.
* Patients providing informed written consent to participate in the study.

Exclusion Criteria:

* Patients with systemic diseases that could influence wound healing (e.g., diabetes, autoimmune disorders).

  * Patients with active periodontal disease.
  * Patients taking medications known to affect bleeding or healing (e.g., anticoagulants, immunosuppressants, steroids).
  * Patients who are pregnant or breastfeeding.
  * Patients who have undergone previous surgical interventions in the palatal donor area.
  * Patients with allergies or hypersensitivity to composite resin materials or collagen-based products.
  * Patients unable or unwilling to comply with postoperative instructions or follow-up visits.
  * Patients with poor oral hygiene or uncontrolled plaque accumulation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | The day of the intervention and every day for the first week
  Measured daily using a Visual Analog Scale (VAS) during the first postoperative week.
General Patient Comfort | The day of the intervention, every day during the first week and 14 days after the intervention
  Evaluated using standardized questionnaires assessing discomfort during daily activities such as eating and oral hygiene
Patient Satisfaction | The day of the intervention, every day during the first week and 14 days after the intervention
  Assessed using Likert scales and validated questionnaires

SECONDARY OUTCOMES:
Clinical Healing of Donor Site | At 7 and 14 days postoperatively.
  Evaluated clinically (e.g., redness, swelling, infection signs) and photographically.
Postoperative Complications | Every day during the first week
  Frequency of events including prolonged bleeding, infection, or need for additional intervention
Analgesic Use | Day of the intervention and every day during the first week.
  Number and duration of analgesic doses prescribed or voluntarily taken by patients
Functional Recovery Time | Every day during the first week and at day 14
  Days required for patients to resume normal activities (e.g., eating without difficulty, returning to work).
Oral Health-Related Quality of Life | At day 14
  Evaluated using standardized questionnaires such as OHIP-14.

CONTACTS AND LOCATIONS:
Locations (1):
- Cagliari University Hospital, Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No